CLINICAL TRIAL: NCT00155610
Title: A Cross-Sectional Study of the Relationship Between Voiding Dysfunction and Intravesical Sensory Threshold in Diabetes Women
Brief Title: The Relationship Between Voiding Dysfunction and Intravesical Sensory Threshold in Diabetes Women
Status: Terminated | Type: Observational
Why Stopped: No clinical significant
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 31MD01
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus
Keywords: diabetic cystopathy; bladder; voiding dysfunction; current perception test
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: intravesical current perception test

SUMMARY:
The investigators will recruit a cross-sectional group of diabetic women in internist clinics. UDS will be applied for voiding function in each case. Intravesical electrical stimulation will be used to test CPT per 5 Hz, 250 Hz, 2000 Hz for the patients. The differences of intravesical CPT between diabetic women with and without voiding dysfunction will be determined.

DETAILED DESCRIPTION:
Diabetes is a common metabolic disease of multiorgan involvement. The American Diabetes Association reported that the prevalence of diagnosed and undiagnosed diabetes mellitus (DM) in the United States is currently 6% and rising. The increase is secondary to a rising incident in obesity, as well as a change in the criteria for the diagnosis of DM from a fasting blood glucose 140 mg/dl to 126 mg/dl. Besides impaired blood glucose regulation, many direct and indirect sequelae of DM can occur. Triopathy of diabetes including retinopathy, neuropathy, and nephropathy are familiar to every internist. Lower urinary tract dysfunction is one of the most common complications in this group of patients.

We look at the difference of intravesical sensation in diabetic women by current perception test; then, we can find the patient with diabetic cystopathy in early stage. We compare the groups of diabetic women with or without voiding dysfunction by urodynamic study. CPT test for intravesical sensation will be applied.

ELIGIBILITY:
Inclusion Criteria:

* The diabetic women followed up in specialist clinics over one year at National Taiwan University Hospital (NTUH)

Exclusion Criteria:

* Concurrent neurological problems or other medical conditions that might interfere with voiding function
* Acute urinary tract infection (UTI)
* Previous pelvic surgery
* Vaginal prolapse

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jeng Yu, MD, Study Chair — Unaffliated